CLINICAL TRIAL: NCT00859352
Title: A Phase I, Open, Randomised, Non-Comparative, Parallel Group Study of a Potential Cytochrome P450 3A Induction After Repeat Twice Daily Oral Dosing With 100 and 500 mg AZD1981 Tablets for 14 Days to Healthy Male Volunteers With Single Oral Doses of Midazolam 7.5 mg.
Brief Title: AZD1981 Midazolam CYP4503A Induction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Christer Hultquist, Medical Science Director, AstraZeneca R&D Lund, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D9831C00008; EudraCT No. 2008-008224-32
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Healthy Male Volunteer
MeSH Terms: interventions — AZD1981; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD1981 100mg and Midazolam
  Interventions: Drug: AZD1981; Drug: Midazolam
- 2 (Experimental): AZD1981 500mg and Midazolam
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: AZD1981 — oral tablets during 14 consecutive days.
  Arms: 1
Drug: Midazolam — Each subject will receive two single doses of 7.5 mg midazolam given as oral solution. The Midazolam dose will be given on Day 1 and on day 16.

SUMMARY:
The primary objective of the study is to investigate if the exposure of midazolam is clinically significantly changed by 14 days of exposure to AZD1981 through possible enzyme induction of CYP3A.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Have a body mass index between 19 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg
* Be a non-smoker or ex-smoker who has stopped smoking for >6 months prior to Visit 1 (pre-entry)

Exclusion Criteria:

* Any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the result of the study, or the subject´s ability to participate
* Any clinically relevant abnormal findings in phys.examination, clinical chemistry, haematology, urinalysis, vital signs, or ECG at baseline which, in the opinion of the investigator, may put the subject at risk because of his participation in the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2009-03; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
PK samples for both AZD1981 and Midazolam. | Intense PK-sampling during 3 pre-defined study days for PK profiling and some sampling throughout the whole study period for confirmatory purposes

SECONDARY OUTCOMES:
Sampling of 4β-hydroxycholesterol | Taken at baseline and after steady state of AZD1981
Safety variables (adverse events and laboratory safety lab) | Adverse events taken during study and safety lab at a few time points

CONTACTS AND LOCATIONS:
Overall Officials: Eva Pettersson, Study Director — AstraZeneca R&D, Lund, Sweden; Aslak Rautio, Principal Investigator — Quintiles Hermelinen AB, Luleå, Sweden
Locations (1):
- Research Site, Uppsala, Sweden